CLINICAL TRIAL: NCT04471298
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Phase 1 Study to Evaluate the Safety and Tolerability of Continuous Oral Treatment With Qishenyiqi Dripping Pills in Healthy Participants
Brief Title: A Study of Qishenyiqi Dripping Pills in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TSL-TCM-QSYQDW-I
Record Dates: First submitted 2020-07-03; First posted 2020-07-15 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Healthy Participants
Keywords: Qishenyiqi Dripping Pills

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Active dosage group 1 (Active Comparator): Qishenyiqi dripping pills, 3.12g, oral, three times a day
  Interventions: Drug: Qishenyiqi dripping pills, 6 bags
- Active dosage group 2 (Active Comparator): Qishenyiqi dripping pills, 4.68g, oral, three times a day
  Interventions: Drug: Qishenyiqi dripping pills, 9 bags
- Active dosage group 3 (Active Comparator): Qishenyiqi dripping pills, 6.24g, oral, three times a day
  Interventions: Drug: Qishenyiqi dripping pills, 12 bags
- Control dosage group 1 (Placebo Comparator): Qishenyiqi dripping pills placebo, 3.12g, oral, three times a day
  Interventions: Drug: Qishenyiqi dripping pills placebo, 6 bags
- Control dosage group 2 (Placebo Comparator): Qishenyiqi dripping pills placebo, 4.68g, oral, three times a day
  Interventions: Drug: Qishenyiqi dripping pills placebo, 9 bags
- Control dosage group 3 (Placebo Comparator): Qishenyiqi dripping pills placebo, 6.24g, oral, three times a day
  Interventions: Drug: Qishenyiqi dripping pills placebo, 12 bags

INTERVENTIONS:
Drug: Qishenyiqi dripping pills, 6 bags — 28 consecutive days
  Arms: Active dosage group 1
Drug: Qishenyiqi dripping pills, 9 bags — 28 consecutive days
  Arms: Active dosage group 2
Drug: Qishenyiqi dripping pills, 12 bags — 28 consecutive days
  Arms: Active dosage group 3
Drug: Qishenyiqi dripping pills placebo, 6 bags — 28 consecutive days
  Arms: Control dosage group 1
Drug: Qishenyiqi dripping pills placebo, 9 bags — 28 consecutive days
  Arms: Control dosage group 2
Drug: Qishenyiqi dripping pills placebo, 12 bags — 28 consecutive days
  Arms: Control dosage group 3

SUMMARY:
This study will evaluate the safety and tolerability of Qishenyiqi Dripping Pills in healthy participants, following oral administration with multiple escalating dose of it.

DETAILED DESCRIPTION:
Qishenyiqi dripping pills, which are made of Huangqi, Danshen, Sanqi, active ingredients of Jiangxiang, have the efficacy of beneficial effects of qi and pulse, blood circulation and pain relief.

This study is a randomized, double-blind, placebo-controlled, dose-escalation design study, including three cohorts and 36 healthy participants. Within each cohort, participant will receive Qishenyiqi dripping pills at the selected dose level by oral administration three times a day for 28 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, male or female, aged 18-50 years (including the boundary value);
* Participants weigh at least 50.0 kg in male and 45.0 kg in female with a body mass index of all subjects between 19 and 26kg/m2 (including the boundary value);
* Participants are willing to have no pregnancy program and take effective contraceptive measures voluntarily since signing informed consent form to 3 months after the last administration;
* Participants are willing to sign Independent Ethics Committee (IEC)-approved informed consent form and able to understand and comply with study procedures.

Exclusion Criteria:

* Participants with allergic constitution or have a history of allergy to drug or food;
* Participants with diseases or physiological conditions that may affect the study, including but not limited to diseases of the nervous, mental, respiratory, cardiovascular, digestive, blood and lymphatic, endocrine, musculoskeletal systems, liver and kidney dysfunction;
* Participants who have any clinically significant abnormalities in vital signs, physical examination, electrocardiogram, chest radiograph, abdominal ultrasound and laboratory examination;
* Participants who have positive test for hepatitis B virus surface antigen (except surface antibodies), hepatitis C virus antibody, human immunodeficiency virus antibody and treponema pallidum antibody;
* Women who are in the state of pregnancy or lactation;
* Participants who have a history of drug abuse or a positive test result for drug abuse at screening;
* Participants who have smoked more than 5 cigarette per day or used a considerable amount of nicotine-containing products within the previous 3 months, and could not quit smoking during the experiment;
* Participants who have been drinking more than 14 units of alcohol per week within the previous 3 months (1 unit ≈285 mL beer with 3.5% alcohol or 25 mL spirits with 40% alcohol or 85 mL wines with 12% alcohol), or positive test for alcohol, or could not abstain from drinking during the trial;
* Participants who have taken any prescription drugs (including prescription, nonprescription, herbal medicine, dietary supplement such as vitamin product and calcium tablet) within 4 weeks before administration of investigational drugs;
* Participants who have difficulty in venous blood collection or history of fainting blood or needles;
* Participants who have participated in any drug clinical trial within 3 months and have taken the experimental drug or plan to participate in other clinical trials during the trial period;
* Participants who have donated or lost blood ≥200 mL within 3 months or received blood transfusion or used blood products, or have blood donation plan during the trial period;
* Judged by the investigator, participants have poor compliance or have other factors such as clinical, social or family that should not be included in the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Adverse events | From screening (2 weeks in advance) till follow-up visit (up to 1week)
  Observe all the adverse events of all participants administrated orally with Qishenyiqi dripping pills.
Number of participants with abnormal vital signs index (body temperature) | From screening (2 weeks in advance) till the end of trial period (Day 29)
  To investigate the safety and tolerability of Qishenyiqi dripping pills following oral administration in healthy participants.
Number of participants with abnormal vital signs index (pulse rate) | From screening (2 weeks in advance) till the end of trial period (Day 29)
  To investigate the safety and tolerability of Qishenyiqi dripping pills following oral administration in healthy participants.
Number of participants with abnormal vital signs index (respiratory rate) | From screening (2 weeks in advance) till the end of trial period (Day 29)
  To investigate the safety and tolerability of Qishenyiqi dripping pills following oral administration in healthy participants.
Number of participants with abnormal vital signs index (blood pressure) | From screening (2 weeks in advance) till the end of trial period (Day 29)
  To investigate the safety and tolerability of Qishenyiqi dripping pills following oral administration in healthy participants.
Physical examination | screening (2 weeks in advance), Day 8, Day 15, Day 22, Day 29
  The complete physical examinations will include an assessment of the general appearance, skin, cardiovascular, abdomen, head, and neck, lymph nodes, musculoskeletal and neurological systems.
Number of participants with abnormal laboratory assessments (blood routine test) | screening (2 weeks in advance), Day 8, Day 15, Day 22, Day 29
  To investigate the safety and tolerability of Qishenyiqi dripping pills following oral administration in healthy participants.
Number of participants with abnormal laboratory assessments (blood biochemical test) | screening (2 weeks in advance), Day 8, Day 15, Day 22, Day 29
  To investigate the safety and tolerability of Qishenyiqi dripping pills following oral administration in healthy participants.
Number of participants with abnormal laboratory assessments (coagulation function test) | screening (2 weeks in advance), Day 8, Day 15, Day 22, Day 29
  To investigate the safety and tolerability of Qishenyiqi dripping pills following oral administration in healthy participants.
Number of participants with abnormal laboratory assessments (urinalysis routine test) | screening (2 weeks in advance), Day 8, Day 15, Day 22, Day 29
  To investigate the safety and tolerability of Qishenyiqi dripping pills following oral administration in healthy participants.
Number of participants with abnormal laboratory assessments (fecal routine test) | screening (2 weeks in advance), Day 8, Day 15, Day 22, Day 29
  To investigate the safety and tolerability of Qishenyiqi dripping pills following oral administration in healthy participants.
Number of participants with abnormal findings in 12-lead safety Electrocardiogram (ECG) | screening (2 weeks in advance), Day 8, Day 15, Day 22, Day 29
  To investigate the safety and tolerability of Qishenyiqi dripping pills following oral administration in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Teaching Hospital of Tianjin University of TCM, Tianjin, Tianjin Municipality, China